CLINICAL TRIAL: NCT05390450
Title: Ultrasound-Guided Popliteal Plexus Block Versus Fascia Iliaca Block for Postoperative Analgesia After Total Knee Arthroplasty: A Randomized Clinical Trial
Brief Title: Ultrasound-Guided Popliteal Plexus Block Versus Fascia Iliaca Block After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Taysser Mahmoud Abdalraheem, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35431/4/22
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Total Knee Arthroplasty; Popliteal Plexus Block; Fascia Iliaca Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Popliteal Plexus Block (Experimental): Patients in this group will receive Popliteal plexus block.
  Interventions: Device: Ultrasound-Guided Popliteal Plexus Block
- Ultrasound-Guided Fascia Iliaca block (Experimental): Patients in this group will receive Fascia Iliaca block.
  Interventions: Device: Ultrasound-Guided Fascia Iliaca block

INTERVENTIONS:
Device: Ultrasound-Guided Popliteal Plexus Block — Patients in this group will receive Popliteal plexus block. Prior to Popliteal plexus block, the proximal end of the adductor canal will be identified. The transducer will be slid distally along the femoral artery until the artery deviated away from the sartorius muscle in the distal part of the adductor canal towards the adductor hiatus. The nerve block needle will be inserted from the anterolateral end of the transducer and advanced in-plane through the medial vastus muscle. The endpoint of injection will be inside the distal end of the adductor canal close to the adductor hiatus. The injection will be adjacent to the femoral artery, between the medial vastus muscle and the adductor magnus muscle. The Popliteal plexus block will be carried out with 10 mL of local anesthetic mixture, containing 50 mg of bupivacaine and 0.05 mg of epinephrine.
  Arms: Ultrasound-Guided Popliteal Plexus Block
Device: Ultrasound-Guided Fascia Iliaca block — Patients will be placed in a supine position, and the skin will be cleaned aseptically. The inguinal ligament from the anterior superior iliac spine to the pubic tubercle will be drawn on the skin and divided into 3 parts. The injection point was 1 cm caudally from the point where the lateral and middle part of the inguinal ligament met. The skin and deep tissues were infiltrated with 1% lidocaine. A 18G nerve block needle will be inserted into the skin perpendicularly until the first (fascia lata) and second loss of resistance (fascia iliaca) will be felt. Following aspiration to exclude intravascular injection, 40 mL of 0.25% bupivacaine (1-1.5 mg/kg), which will be prepared under aseptic conditions, and then injected. Sensorial block will be evaluated using the pinprick test 20 minutes after injection for areas of the thigh innervated by the femoral, lateral cutaneous and obturator nerves.
  Arms: Ultrasound-Guided Fascia Iliaca block

SUMMARY:
This study aims to investigate the effect of the Popliteal Plexus Block versus Fascia Iliaca Block on postoperative pain after total knee arthroplasty.

DETAILED DESCRIPTION:
The Popliteal Plexus entwines the popliteal artery and vein contiguous to the adductor hiatus in the popliteal fossa and innervates the posterior capsule as well as intraarticular genicular structures. It was recently confirmed in a cadaver study that injection of 10 mL of dye into the distal end of the adductor canal spreads via the adductor hiatus to the popliteal fossa and stains the Popliteal Plexus.

Recently, fascia iliaca block was proposed as a popular analgesic technique which involves local infiltration anesthesia under the fascia of the iliacus muscle. The method depends on the local anesthetics spread beneath the fascia to block the peripheral nerve. It has been proposed to avoid the complications by anesthetizing the femoral nerve remotely from major neurovascular structures and achieve adequate analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 75 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) score I-II.
* Scheduled for unilateral, primary TKA under spinal anesthesia.

Exclusion Criteria:

* Coagulopathy.
* Diabetes.
* Obesity.
* Heart failure.
* kidney failure.
* Liver failure.
* Reduced sensation on the lower limb.
* Daily intake of opioids.
* Contraindication to any drug used in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Total intravenous (IV) morphine consumption | 24 hours postoperatively.
  Total intravenous (IV) morphine consumption during the first postoperative 24 hours, postoperatively.

SECONDARY OUTCOMES:
First analgesic request | 24 hours postoperatively
  Time to first analgesic request after surgery in the form of intravenous morphine in a dose (0.05 mg/kg).
Pain level score | 24 hours postoperatively
  Pain levels using the numerical rating scale (NRS) of pain intensity (0 = no pain) to (10 = intolerable pain), pain relief is defined as a NRS of 3 or lower. If the score is >3, the patient will need analgesia in the form of morphine 0.05 mg/kg till it decreases to ≤3. NRS will be assessed and recorded on arrival to Post-Anesthesia Care Unit , 1, 2, 4, 8, 12 and 24 hours postoperatively at rest and on movement (knee flexion) during the first postoperative 24 hours.
Rehabilitation | 24 hours postoperatively
  Rehabilitation (time to ability to sit, time to ability to stand, time to ability to walk, Time to ability to do exercise) will be recorded.
Patient's satisfaction level | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point scale; (1= highly satisfied, 2 = satisfied, 3 = neither satisfied nor unsatisfied, 4 = not satisfied, 5 = highly not satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The protocol will available under reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study.
Access Criteria: The protocol will available under reasonable request from the corresponding author.